CLINICAL TRIAL: NCT00583700
Title: Development of Radiation Fibrosis in Patients Treated With Pentoxyphylline and Vitamin E: a Prospective Randomized Study
Brief Title: Trental & Vitamin E for Radiation-Induced Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200211003
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2012-10

CONDITIONS: Fibrosis
Keywords: Breast Neoplasms; Radiotherapy
MeSH Terms: conditions — Fibrosis; Breast Neoplasms | interventions — Pentoxifylline; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control for study - watchful waiting.
- 2 (Experimental): Combined treatment with Pentoxifylline and Vitamin E.
  Interventions: Drug: Pentoxifylline; Drug: Vitamin E

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400 mg, 3 times daily for 7 months, beginning immediately after radiation therapy.
  Other Names: Trental
  Arms: 2
Drug: Vitamin E — Vitamin E (Over-the-counter) 400 I.U. once daily
  Arms: 2

SUMMARY:
This study seeks to determine if a combination of Trental and Vitamin E prevents the development of radiation fibrosis in women treated with radiation for the definitive management of their breast cancer.

DETAILED DESCRIPTION:
Radiation fibrosis occurs in approximately 25% of those women treated with radiation for breast cancer. Of these, approximately 3 to 5% will develop into an acute, painful form of fibrosis. Mild fibrosis can present as a thicker or more dense breast where the acute form can cause pain in the breast, significant hardening, and inflammation.

Treatments for fibrosis are lacking, with the primary treatment being hyperbaric oxygen therapy. The combination of Trental & Vitamin E has been used with success in Europe and at the University of Iowa.

The focus of this study is to prevent fibrosis through intervention with Trental & Vitamin E. The study has two arms, a control arm and an intervention arm. The study is not blinded. Measurements are taken at standard follow-up visits to measure breast density and lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented cancer of the breast or DCIS or head and neck referred for definitive radiation with curative intent.
* No evidence of metastatic disease.
* Minimum life expectancy of at least 12 months.
* Aged greater than 20 years.
* If female, pregnancy excluded.
* No documented history of collagen vascular disease.

Exclusion Criteria:

* Cognitively impaired patients
* Prisoners
* No histology available
* Documented metastatic disease
* Allergy to Trental
* Life expectance of less than 12 months.
* Aged less than 20 years
* Collagen vascular disease present
* Pregnant
* History of liver disease
* Use of anticoagulants

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-02; Primary Completion 2010-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Jacobson, MD MPH, Principal Investigator — department of radiation oncology
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Dion MW, Hussey DH, Doornbos JF, Vigliotti AP, Wen BC, Anderson B. Preliminary results of a pilot study of pentoxifylline in the treatment of late radiation soft tissue necrosis. Int J Radiat Oncol Biol Phys. 1990 Aug;19(2):401-7. doi: 10.1016/0360-3016(90)90549-y. PMID 2394619
- [Background] Delanian S, Balla-Mekias S, Lefaix JL. Striking regression of chronic radiotherapy damage in a clinical trial of combined pentoxifylline and tocopherol. J Clin Oncol. 1999 Oct;17(10):3283-90. doi: 10.1200/JCO.1999.17.10.3283. PMID 10506631
- [Background] Delanian S, Porcher R, Balla-Mekias S, Lefaix JL. Randomized, placebo-controlled trial of combined pentoxifylline and tocopherol for regression of superficial radiation-induced fibrosis. J Clin Oncol. 2003 Jul 1;21(13):2545-50. doi: 10.1200/JCO.2003.06.064. PMID 12829674
- [Background] Gothard L, Cornes P, Earl J, Hall E, MacLaren J, Mortimer P, Peacock J, Peckitt C, Woods M, Yarnold J. Double-blind placebo-controlled randomised trial of vitamin E and pentoxifylline in patients with chronic arm lymphoedema and fibrosis after surgery and radiotherapy for breast cancer. Radiother Oncol. 2004 Nov;73(2):133-9. doi: 10.1016/j.radonc.2004.09.013. PMID 15542159
- [Background] Delanian S, Porcher R, Rudant J, Lefaix JL. Kinetics of response to long-term treatment combining pentoxifylline and tocopherol in patients with superficial radiation-induced fibrosis. J Clin Oncol. 2005 Dec 1;23(34):8570-9. doi: 10.1200/JCO.2005.02.4729. Epub 2005 Oct 31. PMID 16260695
- See also: Article abstract — http://www.ncbi.nlm.nih.gov/pubmed?term=22846413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2003 and July 2009, 53 breast cancer patients were recruited from the University of Iowa Radiation Oncology clinic and randomized to one of two arms.
Groups:
- Control Arm: Watchful waiting (standard treatment). Study participants received no intervention and were monitored for development of radiation-induced fibrosis.
- Intervention: Pentoxifylline & Vitamin E: Combined treatment with Pentoxifylline and Vitamin E.
  Vitamin E : Vitamin E (Over-the-counter) 400 I.U. once daily
  Pentoxifylline : Pentoxifylline 400 mg, 3 times daily for 7 months, beginning immediately after radiation therapy.
Period: Overall Study
Arm/Group | Control Arm | Intervention: Pentoxifylline & Vitamin E
Started | 27 | 27
Completed | 24 | 23
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention: Pentoxifylline & Vitamin E | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 43
  >=65 years | 2 | 9 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.81) | 59.65 (11.74) | 56.81 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Subjective, Objective, Management, and Analytic (SOMA) Score
Description: A primary outcome of interest is the composite Subjective, Objective, Management, and Analytic (SOMA) score at 18-month follow-up visit. Maximum score is 45, with a score of 0 being ideal and representing no treatment-related side effects at the study visit.
Time Frame: 18 month post-treatment
Population: All participants enrolled in the study were evaluated for SOMA scores. Numbers varied by study participants compliance with follow-up appointments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Arm | Intervention: Pentoxifylline & Vitamin E
Number analyzed (Participants) | 27 | 25
units on a scale | 1.59 (1.53) | 1.0 (1.19)

2. Secondary Outcome: Tissue Compliance
Description: Tissue compliance meter measurements of the treated breast compared to the non-treated breast were obtained at 18 months post-radiation therapy. Tissue compliance simply means how soft and pliable the breast tissue is when force is applied to it.
  One physician would hold the tissue compliance meter (TCM) against the participant's skin. A standard amount of force would be applied. A second physician would read the displacement scale for a specific set of areas on the breast. The range of the scale was 0 to 60 milimeters (mm). The physician's were blineded to the participant's intervention at the time of measurement.
  The final value is the difference between the untreated and the treated breast [untreated - treated]. The range of these differences was -3.3 to 7.0 mm.
Time Frame: 18 months post-treatment
Population: All study participants enrolled were to be measured at 18 months post-radiotherapy. The number of participants analyzed varied by the number compliant with study schedule.
Measure: Mean (Standard Deviation); unit: milimeters (mm)
Arm/Group | Control Arm | Intervention: Pentoxifylline & Vitamin E
Number analyzed (Participants) | 24 | 23
milimeters (mm) | 2.10 (2.16) | 0.88 (1.96)

ADVERSE EVENTS:
Arm/Group | Control Arm | Intervention: Pentoxifylline & Vitamin E
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

LIMITATIONS AND CAVEATS:
Small, single-institutional study. Smaller clinical trials are prone to imbalances in patient characteristics across treatment arms. t tests applied to small studies can be unduly influenced by data that contain outliers or are skewed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes